CLINICAL TRIAL: NCT00209677
Title: Phase I/II Study of Oral S-1 Plus Gemcitabine in Patients With Metastatic Pancreatic Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unfortunately, other Phase III clinical Study (GEM+S-1 vs GEM vs S-1) have been started in Japan.
  h
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Collaborators: Hokkaido University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0405; GEMS-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine
Drug: S-1

SUMMARY:
To assess the usefulness of Gemcitabine plus S-1 therapy based on the antitumor effect and survival period. By performing a phase I/II study of this combination in patients with inoperable or with postoperative pancreatic cancer.

DETAILED DESCRIPTION:
A multicenter Open-label, single-arm, phase I/II clinical trial is conducted on patients with histological stage IV Pancreatic cancer given gemcitabine plus S-1. The usefulness of this regimens as 1st line therapy for pancreatic cancer was evaluated by the disease-free survival(DFS), median survival time (MST), incidence and severity of adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of pancreatic adenocarcinoma.
2. Measurable or assessable lesions(Except for Phase I).
3. Age: 20 ~ 75 years.
4. Kar-nofsky Performance Status (KPS) > 70.
5. No prior chemotherapy
6. No history of treatment with gemcitabine or S-1.
7. No history of radiotherapy to the abdomen.
8. Oral intake of S-1 is possible.
9. Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC 3,500/mm3 and Neutrophil 2,000/mm3. Hb 9.0 g/dl. Platelet count 100,000/mm3. GOT and GPT 2.5 times the upper limit of normal (excluding liver metastasis). T-Bil 2.0 mg/dl. Creatinine within the upper limit of normal). Normal ECG (not considering clinically unimportant arrhythmias and ischemic changes).
10. Predicted survival for >3 months.
11. Able to give written informed consent.

Exclusion Criteria:

1. Severe pleural effusion or ascites.
2. Metastasis to the central nervous system (CNS).
3. Active gastrointestinal bleeding.
4. Active infection.
5. Liver cirrhosis
6. Uncontrolled ischemic heart disease.
7. Serious complications (such as intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, uncontrolled diabetes mellitus, heart failure, renal failure, or hepatic failure).
8. Active multiple cancer.
9. Severe mental disorder.
10. Pregnancy, possible pregnancy, or breast-feeding.
11. Flucytosine treatment
12. Judged to be ineligible for this protocol by the attending physician.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-12; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Determine the DLT(Dose Limiting Toxicity) and MTD(Maximum Tolerated Dose) in Phase I setting.
Determine the clinical response rate with Recommended dose in Phase II setting.

SECONDARY OUTCOMES:
Determine the clinical response rate of patients in Phase I setting.
Determine the MST(Median Survival Time) and DFS(Disease Free Survival) in Phase II setting.

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- Hokkaido University Hospital (Hokkaido University Graduate School of Medicine), Sapporo, Hokkaido, Japan